CLINICAL TRIAL: NCT04667208
Title: Pilot Study: Validation of Easy-to-measure Biomarkers for Intestinal Permeability in Human Trials
Brief Title: Biomarkers for Intestinal Permeability
Status: Completed | Type: Observational
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Prof. Dr., University of Hohenheim
Other Study IDs: Gut barrier study
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Focus: Simplified Method to Assess Intestinal Permeability
Keywords: Gastroenterology; Gut barrier; Intestinal permeability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum and fecal samples will be stored at -80°C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to find easy-to-measure biomarkers of intestinal permeability as surrogate markers for effortful "gold standard" methods.

DETAILED DESCRIPTION:
This study aims to find easy-to-measure biomarkers of intestinal permeability as surrogate markers for effortful "gold standard" methods. In healthy volunteers potential biomarkers for intestinal permeability as well as an established "gold standard" method for intestinal permeability (urinary lactulose/mannitol excretion) will be measured at one time point. Using correlation analyses, potential associations will be assessed and potential biomarkers will be addressed and discussed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written informed consent

Exclusion Criteria:

* Underweight (BMI <18 kg / m2) and obesity from grade II (BMI ≥ 30 kg / m2)
* Acute or chronic gastrointestinal diseases
* Chronically consuming diseases (e.g. chronic tumor disease, florid infections, etc.)
* Smokers (12 hours before the test and during the test it is not allowed to smoke)
* Ingestion of intestinal therapeutics, antibiotics, immunosuppressants or similar within the last 3 months
* Simultaneous participation in another clinical study
* Pregnancy / breastfeeding
* Intolerance to the sugar solution
* Occurrence of relevant diseases
* Revocation of consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Lactulose / mannitol ratio | 1 day (Single measurement)
  Urinary excretion of lactulose and mannitol

SECONDARY OUTCOMES:
Fecal albumin [ng/mg] | 1 day (Single measurement)
  Potential easy-to-measure biomarker #1
Fecal calprotectin [ng/mg] | 1 day (Single measurement)
  Potential easy-to-measure biomarker #2
Fecal zonulin [ng/mg] | 1 day (Single measurement)
  Potential easy-to-measure biomarker #3
Plasma lipopolysaccharide binding protein [µg/ml] | 1 day (Single measurement)
  Potential easy-to-measure biomarker #4

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C Bischoff, Prof. Dr., Principal Investigator — University of Hohenheim, Institute of Nutritional Medicine
Locations (1):
- University of Hohenheim, Stuttgart, Germany